CLINICAL TRIAL: NCT02002442
Title: Comparison of the Effect of the Preoperative Use of Chlorhexidine, Essential Oil, and Cetylpyridinium Chloride Mouthwashes on Bacterial Contamination During Dental Implant Placement: A Randomized Controlled Clinical Trial
Brief Title: Dental Implants and Mouth Rinse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10951
Record Dates: First submitted 2013-11-29; First posted 2013-12-05 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Reduction in Bacterial Counts Through the Use of Mouthwash
Keywords: Mouthwash; Chlorhexidine; cetylpyridinium chloride; Saline; Implants; Saliva Collection
MeSH Terms: interventions — Mouthwashes; Chlorhexidine; Oils, Volatile; Cetylpyridinium; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.12% Chlorhexidine (Active Comparator): Alcohol-free Chlorhexidine Gluconate Oral Rinse USP, 0.12% from GUM®
  Interventions: Other: Mouthwash
- Essential oil (Active Comparator): LISTERINE® ZERO™ Mouthwash
  Interventions: Other: Mouthwash
- 0.07% Cetylpyridinium Chloride (Active Comparator): Crest Pro-Health Multi-Protection Rinse - Refreshing Clean Mint (Procter and Gamble)
  Interventions: Other: Mouthwash
- Saline (Placebo Comparator)
  Interventions: Other: Mouthwash

INTERVENTIONS:
Other: Mouthwash — An investigator will give the patient the assigned mouthwash based on the randomized group allocation. 30ml of the mouthwash will be given to the subject in a sterilized calibrated tube. The subject will be asked to rinse for 60 seconds. Then, the patient will spit the mouthwash.
  Other Names: 0.12% Chlorhexidine; Essential oil; 0.07% Cetylpyridinium Chloride; Saline

SUMMARY:
The primary aim of this study is to evaluate and compare the efficacy of a 60 second rinse with chlorhexidine, essential oil-based mouthwash, cetylpyridinium chloride mouthwash, or saline solution on bacterial contamination in the buccal vestibule when used preoperatively using the real-time Polymerase Chain Reaction (qPCR).

We hypothesize that preoperative rinse with chlorhexidine mouthwash will result in greater reduction of bacterial counts than with essential oil-based, cetylpyridinium chloride, or saline mouthwashes.

The secondary aim of this study is to evaluate the effect of the tested mouthwashes in reducing the bacterial counts over time.

We hypothesize that preoperative rinse with chlorhexidine mouthwash will result in a reduction of bacterial counts for longer duration than with essential oil-based, cetylpyridinium chloride, or saline mouthwashes.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is treatment planned for dental implant placement and qualifies for dental implant placement according to the standards of care in the Department of Periodontology at Tufts University School of Dental Medicine.
* Aged 18 years and above.
* Partially edentulous.

Exclusion Criteria:

* Antibiotic therapy within 2 weeks of the study.
* Active infection in the oral cavity.
* Known allergy to any of the agents used in the study.
* Self-reported pregnancy (as the surgical procedure of dental implant placement is elective and typically deferred until after the delivery).
* Fully edentulous.
* Patient with severe periodontitis (Clinical attachment loss of 5mm or more in the majority of intraoral sites).
* Regular use of mouthwashes (once/day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06

PRIMARY OUTCOMES:
Oral Rinse Comparison | 60 seconds rinse
  The primary aim of this study is to evaluate and compare the efficacy of a 60 second rinse with chlorhexidine, essential oil-based mouthwash, cetylpyridinium chloride mouthwash, or saline solution on bacterial contamination in the buccal vestibule when used preoperatively using the real-time Polymerase Chain Reaction (qPCR).

SECONDARY OUTCOMES:
Bacterial Count Reduction | 60 seconds rinse
  The secondary aim of this study is to evaluate the effect of the tested mouthwashes in reducing the bacterial counts over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University School of Dental Medicine Department of Periodontology, Boston, Massachusetts, United States